CLINICAL TRIAL: NCT04406090
Title: Endovascular Thrombectomy in COVID-19 Infected Patients: Intrahospital and Peri-operative Outcomes
Brief Title: Endovascular Thrombectomy in COVID-19 Infected Patients
Acronym: ET-COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0322
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-05

CONDITIONS: Ischemic Stroke; Covid 19
Keywords: Acute ischemic stroke related to large vessel occlusion; Mechanical Trombectomy; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Ischemic Stroke; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mechanical Trombectomy — Stent retriever for treatment of cerebral arterial occlusions

SUMMARY:
About 5% of COVID-19 patients may present symptoms related to acute ischemic stroke (AIS). Treatment-management and outcomes related to mechanical thrombectomy (MT) for COVID-19 infected patients harboring large vessel occlusion is largely unknown.

This multicentric study aims to investigate morbidity, mortality and neurological outcomes after MT performed in patients with COVID-19 infection.

DETAILED DESCRIPTION:
Since the identification of the first case of Severe Acute Respiratory Syndrome (SARS) CoV-2 infection in December 2019 in Wuhan, China, the global number of confirmed COVID-19 cases is roughly 5 000 000, with 216 involved countries. Increasing evidence shows that SARS-CoV-2 may be associated with neurological manifestations, with up to 36% of patients showing neurological symptoms related to the neurovirulence of the SARS-CoV-2.

It has been reported that roughly 5% of COVID-19 infected patients may present acute ischemic stroke (AIS), and these patients may have an unfavorable clinical evolution due to the systemic involvement of the infective disease. In addition, these patients are quite young: the mean age of COVID-19 patients having AIS is lower (56 years), compared to general population of AIS patients (mean age=73 years). Moreover, most of these patients require an intensive care units (ICU) management. Stroke mechanisms may be multiple and can include hypercoagulability from critical illness, cardioembolism from virus-related cardiac injury, and severe inflammation. Indeed, the dysfunction of endothelial cells induced by infection may promote an increased thrombin generation and fibrinolysis; moreover, the hypoxia found in severe COVID-19 patients can be a trigger for thrombosis, increasing blood viscosity, and inducing hypoxia-inducible transcription factors.

Outcomes related to the treatment of COVID-19 patients harboring large vessel occlusion and requiring MT is substantially unknown, but it is likely that the combined morbidity and mortality rate of the two pathologies is high. Accordingly, patient's selection, treatment-management, and results should be urgently elucidated.

Involving 4 different countries (France, Italy, Spain, and US), this multicentric cohort study aims to analyze the largest possible number of COVID-19 infected patients treated with MT for AIS, with the intention to provide treatment-results and neurological outcomes, elucidating the best patient-selection and treatment-management.

ELIGIBILITY:
Inclusion criteria:

- Patients >18 years infected with the SARR-CoV-2 with acute ischemic stroke, and eligible for mechanical thrombectomy (based on the current guide-lines)

Exclusion criteria:

- Patients <18 years ; no eligibility to mechanical thrombectomy ; absence of diagnosis of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years infected with the SARR-CoV-2, presenting an acute ischemic stroke, and eligible to be treated with mechanical thrombectomy (based on the current guide-lines)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Intrahospital mortality | 1day
  Intrahospital mortality after MT for COVID-19 infected patients harboring large vessel occlusion
short-term morbidity | 1 day
  short-term morbidity after MT for COVID-19 infected patients harboring large vessel occlusion

SECONDARY OUTCOMES:
Angiographic success | 1 day
  Angiographic success after MT for COVID-19 infected patients harboring large vessel occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cagnazzo, MD PhD, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Cagnazzo F, Piotin M, Escalard S, Maier B, Ribo M, Requena M, Pop R, Hasiu A, Gasparotti R, Mardighian D, Piano M, Cervo A, Eker OF, Durous V, Sourour NA, Elhorany M, Zini A, Simonetti L, Marcheselli S, Paolo NN, Houdart E, Guedon A, Ligot N, Mine B, Consoli A, Lapergue B, Cordona Portela P, Urra X, Rodriguez A, Bolognini F, Lebedinsky PA, Pasco-Papon A, Godard S, Marnat G, Sibon I, Limbucci N, Nencini P, Nappini S, Saia V, Caldiera V, Romano D, Frauenfelder G, Gallesio I, Gola G, Menozzi R, Genovese A, Terrana A, Giorgianni A, Cappellari M, Augelli R, Invernizzi P, Pavia M, Lafe E, Cavallini A, Giossi A, Besana M, Valvassori L, Macera A, Castellan L, Salsano G, Di Caterino F, Biondi A, Arquizan C, Lebreuche J, Galvano G, Cannella A, Cosottini M, Lazzarotti G, Guizzardi G, Stecco A, Tassi R, Bracco S, Bianchini E, Micieli C, Pascarella R, Napoli M, Causin F, Desal H, Cotton F, Costalat V; ET-COVID-19 Study Group*. European Multicenter Study of ET-COVID-19. Stroke. 2021 Jan;52(1):31-39. doi: 10.1161/STROKEAHA.120.031514. Epub 2020 Nov 23. PMID 33222617